CLINICAL TRIAL: NCT00000673
Title: A Phase I/II Open-Labelled Trial of Intravitreal Ganciclovir Salvage Therapy for AIDS Patients With Active CMV Retinitis Who Are Intolerant of Systemic Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 085; 11060 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
AMENDED: 04-12-91 Population of patients changed FROM those who are intolerant of systemic therapy with NON-sight-threatening CMV retinitis TO those AIDS patients intolerant of systemic therapy with CMV retinitis.

AMENDED: 8/8/90. Changes made in neutrophils count from < 500 to < 750 cells/mm3. Nonrandomized eyes will not be used for the primary efficacy evaluation.

ORIGINAL DESIGN: To determine the effectiveness and safety of ganciclovir (DHPG) therapy in AIDS patients suffering from active cytomegalovirus (CMV) infection of the retina of the eye (retinitis) when the drug is administered directly into the fluid-filled vitreous cavity of the eye by injection.

CMV retinitis is the most frequently seen opportunistic infection of the eye in AIDS patients, and left untreated can lead to severe visual loss and blindness. While systemic administration of DHPG has been shown to be an effective treatment for CMV retinitis, the chronic administration required may be complicated by decreased blood cell counts (granulocytopenia) which may require discontinuation of treatment. While withholding treatment may allow recovery from the granulocytopenia, interruption of therapy may result in reactivation of the retinitis. Injection of DHPG into the vitreous cavity of the eye may be of benefit to severely neutropenic patients with CMV retinitis.

DETAILED DESCRIPTION:
CMV retinitis is the most frequently seen opportunistic infection of the eye in AIDS patients, and left untreated can lead to severe visual loss and blindness. While systemic administration of DHPG has been shown to be an effective treatment for CMV retinitis, the chronic administration required may be complicated by decreased blood cell counts (granulocytopenia) which may require discontinuation of treatment. While withholding treatment may allow recovery from the granulocytopenia, interruption of therapy may result in reactivation of the retinitis. Injection of DHPG into the vitreous cavity of the eye may be of benefit to severely neutropenic patients with CMV retinitis.

Patients must have active CMV retinitis in one or both eyes, despite prior systemic therapy. Following medical evaluation, the decision is made whether to treat the eye(s) immediately or to watch the eye(s) carefully for advancement of the retinitis. Eyes with sight-threatening lesions or eyes without functional vision are treated immediately and eyes without sight-threatening lesions are randomly chosen for either immediate or deferred therapy. DHPG is given by injection with a very fine needle twice a week for the first 3 weeks and once a week for the remaining 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* AMENDED: 8/8/90 Other available antiretroviral therapy.
* Pneumocystis carinii pneumonia (PCP) prophylaxis, either systemic or local (aerosolized).
* Chemotherapy for Kaposi's sarcoma.
* Systemic therapy for intercurrent opportunistic infections.
* Acyclovir or other treatment of Herpes simplex virus (HSV) or Varicella zoster virus (VZV) infections.
* Systemic therapy deemed necessary for appropriate medical management.

Patients must have AIDS and cytomegalovirus (CMV) retinitis in at least one eye, diagnosed by an ophthalmologist and verified by fundoscopy and fundus photography.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Contraindication to intravitreal injection, including obvious external infection and vitreous hemorrhage.
* Medical opacities of cornea, lens, and/or vitreous which precludes fundus photography.

Concurrent Medication:

Excluded:

* Prophylactic acyclovir at time of study entry.
* Other anticytomegalovirus (CMV) therapy, particularly systemic ganciclovir, foscarnet, or CMV hyperimmune globulin.
* Topical ophthalmic medications should be avoided.
* Cytomegalovirus (CMV) therapies and chronic acyclovir, including necessary therapies for an intercurrent opportunistic infection.

Patients with the following are excluded:

* Contraindication to intravitreal injection, including obvious external infection and vitreous hemorrhage.
* Medical opacities of cornea, lens, and/or vitreous which precludes fundus photography.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Study Completion 1993-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Polsky B, Study Chair
Locations (2):
- United States (2):
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Washington U CRS, St Louis, Missouri

REFERENCES:
- [Background] Polsky B, Wolitz R, Cantrill H, Chuang EL, Heinemann MH, Sands M, Feinberg JE, Power M, Davis R. Intravitreal (IVL) Ganciclovir (GCV) salvage therapy (Rx) for cytomegalovirus (CMV) retinitis (ACTG 085): a preliminary report. Int Conf AIDS. 1991 Jun 16-21;7(2):267 (abstract no WB2340)
- [Background] Polsky, et al. Intravitreal ganciclovir salvage therapy for cytomegalovirus retinitis in AIDS: AIDS Clinical Trials Groups Protocol 085. Int J Infect Dis. 1996 Oct; 1(2):70-4